CLINICAL TRIAL: NCT02259439
Title: Assessment of Updated Evaluation Scores in Critically ILL COPD Patients Admitted to Assiut University Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nermeen Aly Mahmoud Abdel Aleem (Other)
Responsible Party: Sponsor-Investigator, Nermeen Aly Mahmoud Abdel Aleem, chest department- faculity of medicine -Assiut university- Egypt, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 16022012
Record Dates: First submitted 2014-09-17; First posted 2014-10-08 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) represent a leading cause of morbidity and mortality.Patients admitted to hospital present higher mortality rates.The investigators lack the specific tools that allow us to easily classify and establish the individual prognosis for each patient during their hospitalization.

Rational of the study:to identify the predictive factors for hospital mortality in critically ill patients admitted to hospital due to an episode of COPD exacerbation.

DETAILED DESCRIPTION:
Material and Methods:

A) sociodemographic variables:

Age, sex, marital status, occupation, pack\year.

B) clinical variables:

1- Dyspnea measured by the Medical Research Council (MRC) scale and the COPD Assessment Test (CAT ) while stable, previous to admittance.

3- Charlson comorbidity index and age adjusted model.

4- The APACHE II scale: the severity of the episode upon admittance, calculated using the APACHE II scale, using the worst value obtained in the first 24h after being admitted to hospital.

5- the Sequential Organ Failure Assessment (SOFA) scale.

6- Lab parameters: such as glucose, albumin and heamatocrit

7- BAP-65 score: elevated blood urea nitrogen, altered mental status, pulse > 109 beats/min, age > 65 years.

8- Assessment of symptom of gastroesophageal reflux disease.

9-Glasgow scale score.

10-CURB 65 :"C" stands for "confused"; "U" stands for BUN greater than19 mg/dL; "R" stands for "respiration more than 30 breaths per minute""B" stands for blood pressure less than 90 mm Hg systolic or diastolic blood pressure 60 mm Hg or less; "65" stands ≥65 years.

11-CAUDA 70: C: Confusion, Acidosis (pH <7.35), Urea >7mmol/L, MRC Dyspnoea score >4, Albumin <35g/L, Age >70 years. One point was assigned to each variable present, giving a six point scoring system.

12-The COPD and Asthma Physiology Score.

13-The early warning score.

14-ADO index: comprised of age, dyspnea by the MRC, and FEV1. Scores ranged from 0 (best status) to 5 (worst status) for age, 0-3 for MRC, and 0-2 for FEV1. Points for each component were added so that the ADO index ranged from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* We include for study all patients critically ill hospitalized for COPD exacerbation during the study period

Exclusion Criteria:

* Patients who refuse to be admitted to hospital after having been properly informed, and their families as well, of the possible risks that they are assuming.
* Specific diagnosis: pulmonary edema, rib fractures, aspiration, pleural effusion, etc. upon admission.
* Other associated respiratory pathology that determines treatment: pulmonary fibrosis, kyphoscoliosis, neuromuscular pathology, upper airway obstruction, extensive tuberculosis sequelae.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We include for study all patients critically ill hospitalized for COPD exacerbation during the study period.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Calculate the mortality of exacerbated patients based on APACHE II and SOFA score, respiratory rate upon admittance, age, pO2/ FiO2 in the first few hours of admittance. | 24 hours
  Calculate mortality caused by AECOPD depend upon APACHE II and SOFA score

CONTACTS AND LOCATIONS:
Locations (1):
- Chest Department-faculty of medicine-Assuit university, Asyut, Egypt